CLINICAL TRIAL: NCT05564754
Title: Sedation, Temperature and Pressure After Cardiac Arrest and Resuscitation
Acronym: STEPCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University, Lund, Sweden (Unknown); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); The George Institute for Global Health, Australia (Other); HUS Helsinki University Hospitals, Helsinki, Finland (Unknown); Medical Research Institute of New Zealand Rangahautia Te Ora, Wellington, New Zealand (Unknown); University Hospital of Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: step2022
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Arrest With Successful Resuscitation; Hypoxia, Brain
MeSH Terms: conditions — Hypoxia, Brain | interventions — Deep Sedation

STUDY DESIGN:
Intervention Model Description: 2x2x2 factorial, with all patients taking part in each factor.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded. Assessors of neurological prognosis will be blinded. Outcome assessors and investigators will be blinded. Health-care personnel will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Sedation, temperature device and high MAP (Active Comparator): Continuous deep sedation for 36 hours Fever management with a feedback-controlled device if temperature above 37.7°C. A mean arterial pressure target of >85mmHg.
  Interventions: Device: Feedback-controlled temperature device; Other: High MAP; Other: Deep sedation
- Sedation, no temperature device and high MAP (Active Comparator): Continuous deep sedation for 36 hours. Fever management without a feedback-controlled device. A mean arterial pressure target of >85mmHg.
  Interventions: Other: High MAP; Other: Deep sedation; Other: Fever control without a device
- Sedation, temperature device and low MAP (Active Comparator): Continuous deep sedation for 36 hours. Fever management with a feedback-controlled device if temperature above 37.7°C. A mean arterial pressure target of >65mmHg.
  Interventions: Device: Feedback-controlled temperature device; Other: Deep sedation; Other: Low MAP
- Sedation, no temperature device and low MAP (Active Comparator): Continuous deep sedation for 36 hours. Fever management without a feedback-controlled device. A mean arterial pressure target of >65mmHg.
  Interventions: Other: Deep sedation; Other: Fever control without a device; Other: Low MAP
- Minimal sedation, temperature device and high MAP (Active Comparator): Minimal sedation (and early extubation if possible). Fever management with a feedback-controlled device if temperature above 37.7°C. A mean arterial pressure target of >85mmHg.
  Interventions: Device: Feedback-controlled temperature device; Other: High MAP; Other: Minimal sedation
- Minimal sedation, no temperature device and high MAP (Active Comparator): Minimal sedation (and early extubation if possible). Fever management without a feedback-controlled device. A mean arterial pressure target of >65mmHg.
  Interventions: Other: High MAP; Other: Fever control without a device; Other: Minimal sedation
- Minimal sedation, temperature device and low MAP (Active Comparator): Minimal sedation (and early extubation if possible). Fever management with a feedback-controlled device if temperature above 37.7°C. A mean arterial pressure target of >65mmHg.
  Interventions: Device: Feedback-controlled temperature device; Other: Low MAP; Other: Minimal sedation
- Minimal sedation, no temperature device and low MAP (Active Comparator): Minimal sedation (and early extubation if possible). Fever management without a feedback-controlled device. A mean arterial pressure target of >65mmHg.
  Interventions: Other: Fever control without a device; Other: Low MAP; Other: Minimal sedation

INTERVENTIONS:
Device: Feedback-controlled temperature device — If core body temperature exceeds 37.7°C a feedback controlled-device will be used and set at 37.5°C.
  Arms: Minimal sedation, temperature device and high MAP; Minimal sedation, temperature device and low MAP; Sedation, temperature device and high MAP; Sedation, temperature device and low MAP
Other: High MAP — A MAP target of >85mmHg will be used. Vasopressors will be titrated to this target during 36h.
  Arms: Minimal sedation, no temperature device and high MAP; Minimal sedation, temperature device and high MAP; Sedation, no temperature device and high MAP; Sedation, temperature device and high MAP
Other: Deep sedation — Deep sedation for at least 36h
  Arms: Sedation, no temperature device and high MAP; Sedation, no temperature device and low MAP; Sedation, temperature device and high MAP; Sedation, temperature device and low MAP
Other: Fever control without a device — Management of fever in the ICU without a device
  Arms: Minimal sedation, no temperature device and high MAP; Minimal sedation, no temperature device and low MAP; Sedation, no temperature device and high MAP; Sedation, no temperature device and low MAP
Other: Low MAP — A MAP target of >65mmHg will be used. Vasopressors will be titrated to this target during 36h.
  Arms: Minimal sedation, no temperature device and low MAP; Minimal sedation, temperature device and low MAP; Sedation, no temperature device and low MAP; Sedation, temperature device and low MAP
Other: Minimal sedation — A strategy of minimal sedation in the ICU, used only as needed to facilitate transport, imaging and invasive procedures.
  Arms: Minimal sedation, no temperature device and high MAP; Minimal sedation, no temperature device and low MAP; Minimal sedation, temperature device and high MAP; Minimal sedation, temperature device and low MAP

SUMMARY:
The STEPCARE-trial is a 2x2x2 randomised trial studying patients who have been resuscitated from cardiac arrest and who are comatose. It will include three different interventions focusing on sedation targets, temperature targets and mean arterial pressure targets.

DETAILED DESCRIPTION:
3500 patients who are comatose after cardiac arrest will be included in a trial studying three separate targets. All patients will be randomised to a control or an intervention arm for sedation, temperature and blood pressure targets. These are.

1. Continuous deep sedation for 36 hours or minimal sedation (SEDCARE)
2. Fever management with or without a feedback-controlled device (TEMPCARE)
3. A mean arterial pressure target of >85mmHg or >65mmHg. (MAPCARE)

Participants will be followed up at 30 days and 6 months. The primary outcome will be survival at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Out-of-hospital cardiac arrest
2. Sustained ROSC - defined as 20 minutes with signs of circulation without the need for chest compressions
3. Unconsciousness defined as not being able to obey verbal commands (FOUR-score motor response of <4) or being intubated and sedated because of agitation after sustained ROSC.
4. Eligible for intensive care without restrictions or limitations
5. Inclusion within 4 hours of ROSC

Exclusion Criteria:

1. On ECMO prior to randomization
2. Pregnancy
3. Suspected or confirmed intracranial hemorrhage
4. Previously randomized in the STEPCARE trial
5. Trauma or hemorrhage being the presumed cause of arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 6 months
  Landmark mortality at follow-up performed at 6 months

SECONDARY OUTCOMES:
Functional outcome | 6 months
  Proportion of patients who have a mRS score of 4-6
Health-related quality of life | 6 months
  EQ5D-5L VAS

OTHER OUTCOMES:
ICU stay | 6 months
  Length of stay for ICU survivors
Days at home within the first 30 days | 30 days
  Days outside of hospital within the first 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Nielsen, PhD, Study Chair — Lund University
Locations (56):
- Australia (8):
  - Nepean Hospital, Kingswood, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - The Sutherland Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - The Prince Charles Hospital, Brisbane, Queensland
  - Austin Hospital, Melbourne, Victoria
- Belgium (3):
  - HUB Hôpital Erasme, Brussels
  - Ghent University Hospital, Ghent
  - Ziekenhuis Oost-Limburg Hospital, Lanaken
- North Estonia Medical Centre, Tallinn, Tallinn, Estonia
- Finland (7):
  - Jorvi Hospital, Espoo
  - Meilahti Hospital, Helsinki
  - Helsinki Helsingforgs University Central Hospital, Helsinki
  - Jyväskylä Hospital, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
- Germany (3):
  - Charite University Hospital, Berlin
  - Lübeck University Hospital, Lübeck
  - Tubingen University Hospital, Tübingen
- St Vincents University Hospital, Dublin, Ireland
- San Martino Hospital Genova, Genova, Italy
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- New Zealand (6):
  - DCCM ICU, Auckland
  - Middlemore ICU, Auckland
  - North Shore ICU NZ, Auckland
  - Christchurch Hospital, Christchurch
  - Whangarei ICU, Northland
  - Wellington Hospital, Wellington
- Norway (4):
  - Soerlandet Hospital Arendal, Arendal
  - Kalnes Hospital, Kalnes
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
- King Abdulaziz Medical City, Riyadh, Saudi Arabia
- Tan Tock Seng Hospital, Singapore, Singapore
- Sweden (9):
  - Hallands hospital, Halmstad, Halland County
  - Helsingborg Hospital, Helsingborg, Skåne County
  - Skåne University Hospital, Lund, Skåne County
  - Skåne University Hospital Malmö, Malmo, Skåne County
  - Sahlgrenska University Hospital, Gothenburg
  - Karlstad hospital, Karlstad
  - Skaraborg Hospital Skovde, Skövde
  - Karolinska University Hospital, Stockholm
  - University Hospital of Umeå, Umeå
- Switzerland (3):
  - Bern University Hospital, Bern
  - St Gallen Hospital, Sankt Gallen
  - University Hospital Zürich, Zurich
- United Kingdom (7):
  - Essex Cardiothoracic Centre, Basildon
  - Bristol Royal Infirmary, Bristol
  - Cardiff University Hospital, Cardiff
  - Leeds General Infirmary, Leeds
  - Kings College Hospital, London
  - St Bartholomew's Hospital, London
  - St Georges University Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request following publication

REFERENCES:
- See also: Trial webpage — http://stepcare.org